CLINICAL TRIAL: NCT06320990
Title: A Pilot Study of Chemoprevention With Tamoxifen in Patients With Pre-Invasive Pancreas Mucinous Cystic Neoplasms Who Will Not Undergo Immediate Resection
Brief Title: Chemoprevention With Tamoxifen in Pre-Invasive Pancreas Mucinous Cystic Neoplasms Not Undergoing Immediate Resection
Acronym: MCN_Tam
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0074-24-CB
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Pancreatic Cyst; Pancreatic Mucinous Cystic Neoplasm
MeSH Terms: conditions — Pancreatic Cyst | interventions — Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tamoxifen (Experimental): Tamoxifen 20mg by mouth daily for up to 6 months
  Interventions: Drug: Tamoxifen 20mg

INTERVENTIONS:
Drug: Tamoxifen 20mg — Tamoxifen is a nonsteroidal antiestrogen for oral administration.
  Other Names: Soltamox

SUMMARY:
Pancreatic mucinous cystic neoplasm (MCN) is a precursor to invasive pancreatic adenocarcinoma which occurs almost exclusively in females in their 5th-7th decade. Currently the only option for MCN treatment and prevention of invasive pancreatic ductal adenocarcinoma (PDA) is oncologic resection. The clinical features of pancreatic MCN support the influence of sex hormones in the pathogenesis of the disease. Anti-hormonal therapy may therefore constitute an effective approach to treatment. Preliminary analyses from preclinical studies suggest that tamoxifen inhibits the spread and normal life cycle in MCN epithelial cells and fibroblasts. Investigators hypothesize that in humans, treatment with tamoxifen will lead to cyst regression or stabilization and may spare or delay the need for resection. Up to 15 participants not undergoing immediate resection will be enrolled and take tamoxifen orally for up to 24 weeks. The study will assess the feasibility of tamoxifen as a treatment for pancreatic MCN.

DETAILED DESCRIPTION:
Pancreatic mucinous cystic neoplasm (MCN) is a precursor to invasive pancreatic adenocarcinoma which occurs almost exclusively in females in their 5th-7th decade. Currently the only option for MCN treatment and prevention of invasive pancreatic ductal adenocarcinoma (PDA) is oncologic resection. The clinical features of pancreatic MCN support the influence of sex hormones in the pathogenesis of the disease. Anti-hormonal therapy may therefore constitute an effective approach to treatment. Preliminary analyses from pre-clinical studies suggest that tamoxifen inhibits proliferation and apoptosis in MCN epithelial cells and fibroblasts. Investigators hypothesize that in humans, treatment with tamoxifen will lead to cyst regression or stabilization and may spare or delay the need for resection.

This is an open-label pilot study of tamoxifen as chemoprevention in participants with pancreatic mucinous cystic neoplasms (MCN) who will not undergo immediate resection. Up to 15 participants will be enrolled and take tamoxifen 20mg by mouth daily for up to 24 weeks. The study will assess the feasibility of tamoxifen as chemoprevention in participants with pancreatic MCN and objective response rate as assessed by magnetic resonance imaging (MRI). This study is intended to inform the design of a subsequent trial formally powered to detect the benefit of tamoxifen in treating pancreatic MCN.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 19 years
* Clinically diagnosed pre-invasive pancreatic mucinous cystic neoplasm (MCN), measurable by cross-sectional imaging
* Surgical resection of the lesion is not planned due to cyst features, patient factors or patient preference
* Females of reproductive potential and males with partners of reproductive potential must agree to employ two methods contraception throughout the study and for up to 3 months following treatment. Non-child-bearing potential is defined as age 45 years or older and no menses for greater than or equal to 12 months or any age with surgical removal of the uterus and/or both ovaries.
* Estimated glomerular filtration rate (eGFR) > 30mL/min/1.73m2
* Willing and able to provide informed consent to and abide by the protocol

Exclusion Criteria:

* Presence of invasive pancreatic adenocarcinoma or high-grade dysplasia
* Presence of a solid component or mural nodule, main pancreatic duct dilation or abrupt caliber change, obstructive jaundice, lymphadenopathy
* Current or prior use of tamoxifen or another estrogen antagonist including, but not limited to, clomifene, raloxifene, fulvestrant, anastrazole; subjects who have previously used an estrogen antagonist are eligible provided the last use was at least 5 years prior to enrollment.
* Current or planned use of hormonal treatments including estrogen, progesterone, androgens, hormone replacement therapy or other types of hormonal contraceptives including implants and depot injections; levonorgestrel-releasing intrauterine device (IUD) is permitted.
* Contraindications to tamoxifen include:

  * Pregnancy or nursing
  * Known allergy or hypersensitivity to tamoxifen
  * Cataracts which affect visual acuity (ie. symptomatic)
  * Retinopathy which affects visual acuity (ie. symptomatic)
  * Current warfarin use
  * History of deep vein thrombosis or pulmonary embolism or other condition which, in the opinion of the investigator, may significantly increase the individual's risk of venous thromboembolism
  * History of stroke
  * Known endometrial hyperplasia or personal history of endometrial carcinoma, uterine sarcoma and uterine carcinosarcoma
* History of intestinal disease or major gastric surgery likely to alter absorption of tamoxifen or inability to swallow oral medications
* Uncontrolled illness including but not limited to ongoing or active infection requiring IV antibiotics, symptomatic congestive heart failure, unstable angina or uncontrolled cardiac arrhythmias, or other conditions which might jeopardize or preclude the ability of the patient to take tamoxifen or the safety of follow-up visits, scans and procedures
* Elective surgery planned for the study period
* Participation in another clinical study with an investigational product during the last 28 days
* Any participant, in the opinion of the investigator, who will not be able to tolerate treatment, or the participant is unsuitable to participate in the study and is unlikely to comply with study procedures, restrictions and requirements

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Feasibility, by adherence rate | 6 months (approximately 180 days)
  Adherence rate, defined as the proportion of participants who take ≥70% of the prescribed tamoxifen doses with adherence at least 60%, meaning ≥60% of participants take ≥70% of the prescribed tamoxifen doses.
Feasibility, by retention rate | 6 months (approximately 180 days)
  Retention rate, defined as the proportion of participants who complete imaging and study procedures at the 6-month visit with retention of at least 50%, meaning at least 50% of participants complete imaging and study procedures at the 6-month visit.

SECONDARY OUTCOMES:
Objective response rate (ORR) of pancreatic MCN | 12 months (approximately 360 days)
  The ORR will be estimated based on the proportion of participants with complete or partial response on MRI/MRCP; partial response is defined by ≥ 20% decrease in maximal cyst diameter.

CONTACTS AND LOCATIONS:
Overall Officials: Kelsey Klute, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No